CLINICAL TRIAL: NCT07233356
Title: Novel Risk Factors and Localization of Peripheral Arterial Disease
Acronym: GWADAOMI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RI2_2017/10
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Atherosclerotic Peripheral Arterial Disease; Hemoglobin A1c Protein, Human; Guadeloupe
Keywords: Hemoglobin A1c; Atherosclerotic peripheral arterial disease; distal localization,; novel risk factors,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood and urinary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: culprit lesion is infra popliteal
- group 2: culprit lesion is supra or popliteal

SUMMARY:
Background: .Atherosclerotic peripheral arterial disease (PAD) is associated with a high risk of mortality, coronary events and stroke. The distal localization is frequently associated with amputation. Patients from African origin have a higher prevalence of PAD independently of age and other risk factors. In Guadeloupe, French West Indies, infra popliteal localization is more frequent than in France continental associated with different risk factors (88% of hypertension, 2/3 of diabetes).

Purpose: Traditional risk factors of PAD are smoking diabetes, hypertension, high lipid levels, age, and family history of cardiovascular events. The role of novel risk factors in PAD has recently been shown: fibrinogen, CRP-us, homocysteine, interleukin 6, the neutrophil-to-lymphocyte ratio, the urinary albumin-to-creatinine ratio, alkaline phosphatases, insulin resistance, uric acid, D dimer, vitamin D deficiency, HBA1C. Thus the purpose of the research is to study the role of novel risk factors in the occurrence of infrapopliteal PAD. The primary criterion is the HBA1C.

DETAILED DESCRIPTION:
In Guadeloupe, French West Indies, a high prevalence of distal (infra popliteal) PAD has been observed compared to France continental, the risk factors associated with the distal localization are diabetes and hypertension. Novel risk factors in PAD have been highlighted such as fibrinogen, CRP-us, homocysteine, interleukin 6, the neutrophil-to-lymphocyte ratio, the urinary albumin-to-creatinine ratio, alkaline phosphatases, insulin resistance, uric acid, D dimer, vitamin D deficiency. HBA1 C is also an independent novel risk factor of PAD in diabetic and non-diabetic patients. It seems that risk factors are different according to the localization of the disease. Thus the aim of the research is to study the role of novel risk factors in the localization of PAD. The primary outcome is the HBA1C. The secondary outcome is the role of other risk factors in the localization of PAD. This is a cross sectional study. Patients with PAD diagnosed with systolic pressure index< 0.9 or toe systolic pressure < 85 mmHg or tissue oxygen saturation <65 mmHg or with stenosis > 50 % or occlusion will be proposed to participate in the study. If the culprit lesion is infra popliteal they will be included in group 1. If the culprit lesion is supra or popliteal they will be included in group 2. Patients will be informed of the study and the written informed consent will be obtained. Clinical and para clinical date will be taken on the same date (V0). Then the patient will have to go to the Pointe à Pitre hospital within one month for a second visit (V1) where blood and urinary samples will be taken. Interleukin 6 and insulin in non-diabetic and blood collection will specially be taken for the study.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged more than 18 years old
* with PAD diagnosed with systolic pressure index (SPI) <0.9 or toe systolic pressure <85 mmHg or tissue oxygen saturation < 65 mmHg or with stenosis >50 % or occlusion of one or more arteries
* Patients with or without diabetes
* with stenosis >50 % or occlusion of one or more arteries, infra popliteal, supra or popliteal
* wishing to take part in the study
* having signed the informed consent
* Patients affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Patients aged less than 18 years old
* Patients who do not wish to participate in the study
* Patients with PAD with localization infra popliteal and supra popliteal or popliteal (stenosis > 50 % or occlusion of an artery at supra popliteal or popliteal level AND infra popliteal level)
* Patients with an history of revascularization at supra popliteal, popliteal or infra popliteal level AND stenosis on a different territory.
* Patients with medial calcific sclerosis without PAD
* PAD from non-atherosclerotic origin
* Patient non-affiliated to the social security scheme
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a Doppler ultra sound for known PAD or newly diagnosed PAD at hospital or at vascular doctor's offices will be proposed to participate in the study. PAD will be diagnosed if systolic pressure index< 0.9 or toe systolic pressure < 85 mmHg or tissue oxygen saturation <65 mmHg or if there is a stenosis > 50 % or an occlusion.. If the culprit lesion is infra popliteal they will be included in group 1. If the culprit lesion is supra or popliteal they will be included in group 2.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | between day 0 to month 3
  pourcentage

SECONDARY OUTCOMES:
novel risk factors fibrinogen | between day 0 and month 3
  g/L
novel risk factors homocysteine | between day 0 an month 3
  umol/L
novel risk factors interleukin 6, | between day 0 and month 3
  pg/mL
novel risk factors neutrophil-to-lymphocyte ratio, | between day 0 and month 3
  value
novel risk factors urinary albumin-to-creatinine ratio | between day 0 and month 3
  mg/g
novel risk factors alkaline phosphatases, | between day 0 and month 3
  U/L
novel risk factors insulin resistance, | between Day 0 and month 3
  value
novel risk factors uric acid, | between day 0 and month 3
  umol/L
novel risk factors D dimer | between day 0 and month 3
  ng/mL
novel risk factors vitamin D deficiency. | between day 0 and month 3
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Anne BLANCHET, Doctor, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Centre Hospitalier Universitaire de la Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe